CLINICAL TRIAL: NCT06316661
Title: MAgnetic Resonance Non-contrast Assessment of Cardiac Microvascular Dysfunction in Patients With Heart Failure With PrEserveD Ejection Fraction (MAPPED)
Brief Title: CMR Assessment of Cardiac Microvascular Dysfunction in Patients With HFpEF
Acronym: MAPPED
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09C921
Record Dates: First submitted 2024-03-05; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Microvascular Coronary Artery Disease; Heart Failure With Reduced Ejection Fraction
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HFpEF: patients with HFpEF
  Interventions: Diagnostic Test: stress perfusion cardiac magnetic resonance; Diagnostic Test: cardiopulmonary exercise test
- healthy volunteers: healthy volunteers matched for age and sex
  Interventions: Diagnostic Test: stress perfusion cardiac magnetic resonance; Diagnostic Test: cardiopulmonary exercise test

INTERVENTIONS:
Diagnostic Test: stress perfusion cardiac magnetic resonance — stress perfusion cardiac magnetic resonance according to guidelines, with quantitative evaluation for microvascular dysfunction assessment
Diagnostic Test: cardiopulmonary exercise test — bike exercise with ECG and non invasive respiratory gas exchange monitoring

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) causes hospitalizations, premature mortality and high health care costs. This is also due to poor understanding of HFpEF pathogenesis and, thus, lack of specific therapies. Prompted by the recent demonstration that HFpEF clusters different clinical phenotypes, the investigators propose that these phenogroups are driven by distinct myocardial abnormalities. Cardiac Magnetic Resonance (CMR) can help filling this gap in knowledge: on top of providing gold standard measurements for myocardial volume and cellular mass, recent technical advantages mean that this test can assess and quantify left ventricular extracellular volume, fibrosis and microvascular function accurately and non-invasively. In HFpEF patients, the investigators aim at assessing 1) the coronary microvascular function impairment; 2) the myocardial fibrotic burden; - seeking to understand the disease in order to improve care and cardiovascular outcomes for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age greater of or equal to 18 years at enrolment
* Able to provide written informed consent
* Diagnosis of HFpEF as defined by the 2016 ESC Guidelines (only for HFpEF group)

Exclusion Criteria:

* Pregnancy or breastfeeding
* Absolute contraindication to adenosine perfusion cardiac MRI (including uncontrolled asthma and severe chronic kidney failure, defined as glomerular filtration rate < 30ml(min/kg)
* Atrial fibrillation
* Previous chemotherapy and/or mediastinal radiotherapy
* Known CAD
* Diabetes Mellitus
* Systemic inflammatory diseases
* Any other medical condition which, in the Investigators' opinion, could affect the study results
* Only for control group: any known cardiac, pulmonary, haematological or neoplastic known medical condition and/or any chronic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: N=40 patients will be recruited in the HFpEF group (from now on "HFpEF"), N=20 in the control group (from now on "Controls").
  * HFpEF: Eligible HFpEF patients will be identified in the Auxologico Outpatient Clinics (in particular in the Dyspnoea and Pulmonary Hypertension Clinic, run by Dr Sergio Caravita), with the aim to include 20 patients with early stages of disease (high filling pressure only during exercise, with nonconclusive results of rest examinations, roughly corresponding to Shah's phenogroup n 1) and 20 patients with advanced stages of disease (signs of pulmonary hypertension and right ventricular dysfunction, roughly corresponding to Shah's phenogroup n 3).
  * Controls: healthy volunteers will be matched for age and gender to the HFpEF.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Peak stress perfusion | at recruitment (cross sectional)
  Detection of impaired cardiac microvascular function (defined as a T1 mapping reactivity - delta T1m before and during stress test= 3.0 +/-0.9%) in HFpEF patients compared to healthy controls.
Extracellular volume | at recruitment (cross sectional)
  Detection of higher cardiac diffuse fibrosis (defined as increased extracellular volume, measured by T1 mapping as per international guidelines, expressed as % ) in HFpEF patients compared to healthy controls.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Auxologico Italiano, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes